CLINICAL TRIAL: NCT00525577
Title: AGI-1067 as a Novel Antidiabetic Agent Evaluation Study
Brief Title: ANDES-AGI-1067 as a Novel Antidiabetic Agent Evaluation Study
Acronym: ANDES
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: AtheroGenics (Industry)
Responsible Party: Walker Long, MD, AtheroGenics, Inc
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AGI-1067-052
Record Dates: First submitted 2007-09-04; First posted 2007-09-06 (Estimated); Last update posted 2008-02-06 (Estimated); Status verified 2008-02

CONDITIONS: Diabetes
Keywords: Type 2 diabetes, glycemic control
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — succinobucol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1:A (Experimental): Placebo
  Interventions: Drug: Placebo
- 2:B (Experimental): AGI-1067 75 mg
  Interventions: Drug: AGI-1067
- 3:C (Experimental): AGI-1067 150 mg
  Interventions: Drug: AGI-1067

INTERVENTIONS:
Drug: Placebo — Placebo tablet, once daily
  Arms: 1:A
Drug: AGI-1067 — 75 mg AGI-1067 tablet, once daily
  Other Names: AGI-1067 (succinobucol)
  Arms: 2:B
Drug: AGI-1067 — 150 mg AGI-1067 Tablet, once daily
  Other Names: AGI-1067 (succinobucol)
  Arms: 3:C

SUMMARY:
This double-blind, placebo-controlled, dose-finding study is designed to identify the lowest AGI-1067 dose that improves glycemic control as measured by HbA1c and fasting glucose in subjects with Type 2 diabetes mellitus. Glycemic control will be measured during a 6-month treatment period in subjects who are on 1 or no antidiabetic drugs

ELIGIBILITY:
Inclusion Criteria:

1. Provide informed written consent prior to entry.
2. Be male or female 18-75 years of age at the time of entry and have Type 2 diabetes for a minimum of 6 months prior to Screening 1 visit.
3. Have an HbA1c level measured at the Screening 1 and Screening 2 visits with a minimum level at ≥7.5% for both visits, as determined by the core lab analysis.
4. Be taking either 1 or no antidiabetic agents. If on an antidiabetic medication, it must be of the sulphonylurea, metformin, or glitazone class, and the dosage must have been stable for the last 3 months prior to the Screening 1 visit. Note that no combination medications (i.e., counted as more than 1 agent) will be permitted prior to Randomization and that the use of GLP mimetrics, DPPIV inhibitors, or colesevelam are not permitted (rescue medication will be allowed at 3 months).
5. Subjects who are using hormone replacement therapy must have been on stable doses of their hormone replacement therapy for at least 3 months prior to the Screening 1 visit.
6. Females must not be breast feeding or pregnant. If they are of child-bearing potential, they must be using a reliable method of birth control considered suitable by the Investigator. If on hormonal contraceptives for more than 6 months, subjects will be allowed to participate in the study provided that this therapy remains constant throughout the study and for a period of 2 months after the end of the study.

Exclusion Criteria:

1. Have Type 1 diabetes or history of ketoacidosis determined by medical history
2. Have an HbA1c of more than 10.5% or a fasting glucose of >240 mg/dL (13.3 mmol/L) at either the Screening 1 [Visit 1] or Screening 2 [Visit 2])
3. Have a history of severe diabetic neuropathy including autonomic neuropathy, gastroparesis, or lower limb ulceration or amputation.
4. Have a history of long-term therapy with insulin (>30 days) within the last year or >7 days within the last 3 months.
5. Require parenteral corticosteroids or recurrent continuous oral corticosteroid treatment (>2 weeks) within the last 3 months.
6. Use weight loss drugs (e.g., orlistat, sibutramine, phenylpropanolamine, phentermine, or similar prescription or over-the-counter medications) within 3 months of the Screening 1 visit or intentional weight loss of ≥4 kg in the previous 6 months.
7. Have had a new antidiabetic medication added, or the dose of an existing antidiabetic medication changed, in the last 3 months prior to the Screening 1 visit.
8. Have had a stroke, MI, coronary artery bypass graft (CABG), percutaneous transluminal coronary angioplasty (PTCA), or admission with unstable angina within the last 6 months prior to the Screening 1 visit.
9. Have congestive heart failure New York Heart Association Class III or IV (Appendix B).
10. Have taken any of the following drugs in 6 months prior to the Screening 1 visit: cholestyramine, colestid, cyclosporine, or isotretinoin.
11. Have acute infections requiring parenteral antibiotic treatment within the last 3 months.
12. Have uncontrolled hypertension (defined as systolic blood pressure >180 mmHg).
13. Have platelets <100,000 K/cu mm (x 103/μL) at the Screening 1 visit.
14. Have active liver disease or hepatic dysfunction (total bilirubin, aspartate aminotransferase [AST], alanine aminotransferase [ALT] >1.5 times upper limit of normal [ULN]) as determined by core lab analysis at either the Screening 1 visit or the Screening 2 visits.
15. Subjects with long QT syndrome as evidence by a QTc at the Screening 1 visit of >460 msec in males or >480 msec in females or subjects taking and requiring continued therapy with antiarrhythmic medications such as sotalol, quinidine, dofetilide, amiodarone or other drugs known to significantly prolong the QT interval (this will not include drugs associated with minor effect on the QT interval of less than 15 msec.)
16. Have known major chronic infection or major hematologic, renal, metabolic, gastrointestinal or endocrine dysfunction in the judgment of the Investigator (including diabetes mellitus too severe to allow the subject to safely participate in this study).
17. Have had a life-threatening illness or any history of cancer or malignancy within the past 5 years (except for basal cell carcinoma).
18. Have had surgery requiring inpatient admission within 30 days prior to the Screening 1 visit.
19. Considered unreliable as a study participant based on the Investigator's (or designee's) knowledge of the subject (e.g., history of alcohol or other drug abuse, inability or unwillingness to adhere to the protocol, or psychosis).
20. Have a history of intolerance or previous use of probucol within the last 5 years.
21. Have participated in a previous study with AGI-1067.
22. Have participated in any investigational drug study within 30 days prior to study entry, or expects to participate in any other investigational drug study during the course of ANDES.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1012 (Estimated)
Dates: Start 2007-08; Primary Completion 2008-06 (Estimated); Study Completion 2008-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in HbA1c to the 6-month time point is identical in the study groups (placebo and AGI-1067 treatment groups) | 6 month

SECONDARY OUTCOMES:
• Change of HbA1c from baseline throughout the study • Change of FPG from baseline throughout the study• | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Walker Long, MD, Study Chair — AtheroGenics, Inc
Locations (90):
- United States (2):
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Diabetes and Glandular Disease, San Antonio, Texas
- Clinic for the Internal Medicine-Clinical Center Banja Luka, Banja Luka, Bosnia and Herzegovina
- Georgia (7):
  - Center of Endocrinology, Metabology & Nutriology, Tbilisi
  - Diagnostic Services Ltd., Tbilisi
  - Georgian Diabetes Center, Tbilisi
  - Healthy Life Center, Tbilisi
  - Institute of Cardiology, Tbilisi
  - Tbilisi Center of Endocrinology, Tbilisi
  - Tbilisi State Medical University Clinic #1, Tbilisi
- India (30):
  - Second floor , Silver Brook Building,, Ahmedabad
  - Shantiniketan Hospital, Ahmedabad
  - Bangalore Diabetes, Bangalore
  - Bhagwan Mahaveer Jain Hospital, Bangalore
  - M.s. Ramaiah Memorial Hospital, Bangalore
  - St. Johns Medical College and Hospital,, Bangalore
  - Belgaum Diabetes Centre, Belagavi
  - Dr. V Seshiah Diabetes Care and Research Institute, Chennai
  - Madras Research Center, Chennai
  - Sri Ramachandra Medical Centre, Chennai
  - Mediciti Hospital, 5-9-22, Hyderabaad
  - Medwin Hospitals, Hyderabaad
  - Sai's Endocrine and Growth Centre, Hyderabaad
  - Diabetes, Thyroid and Endocrine, Jaipur
  - Saytam Hospital and Research Centre, Jaipur
  - Amrita Institute of Medical Sciences, Kochi
  - Dayanand Medical College & Hospital, Ludhiana
  - IRL-Synexus Clinical Research Centre, Mumbai
  - Medicine C Railway Hospital, Byculla, Mumbai
  - T.N.M. College & BYL Nair CH, Mumbai
  - TMMC&LTMGH, Sion Hospital, Mumbai
  - All India Institute of Medical Sciences, New Dehli
  - Apollo Health Education Research and Foundation(AHERF), New Dehli
  - Fortis Flt. Lt. Rajan Dhall Hospital, New Dehli
  - Maulana Azad Medical College and Lok Nayak Hospital, New Dehli
  - Sir Ganga Ram Hospital, New Dehli
  - Jehangir Hospital, Pune
  - Orange Diabetes Speciality Clinic, Pune
  - SUT Hospital, Trivandrum
  - Endocrine & Diabetes Centre, Visakhapatnam
- North Macedonia (4):
  - Clinical Hospital "Dr. Trifun Panovski", Bitola
  - General Hospital, Kumanovo, Kumanovo
  - General Hospital, Ohrid,, Ohrid
  - University Clinical Center Skopje, Skopje
- Serbia and Montenegro (6):
  - Institute for Endocrinology, Diabetes and Metabolic-Clinical Center Serbia, Belgrade
  - Clinic for the Internal Medicine-Clinical Cente Bijelo Polje, Bijelo Polje
  - Clinic for the Internal Medicine-Clinical Cente Kotor, Kotor
  - Clinic for the Internal Medicine-Clinical Cente Kragujevac, Kragujevac
  - Clinic of endocrinologyClinical Center Nis, Nis
  - Clinic for the Internal Medicine-Clinical Center Podgorica, Podgorica
- South Africa (27):
  - Josha Research, Rubins Building, Bloemfontein
  - Quinta Research, Bloemfontein
  - 21 Concert Boulevard, Cape Town
  - Brooklyn Medical Centre, Cape Town
  - Paarl Research Centre, Medicross Paarl, Cape Town
  - Tiervlei Trial Centre, Karl Bremer Hospital, Cape Town
  - TREAD Research Tygerberg Hosp, Cape Town
  - 8 Flamco Terrace, Chatsworth
  - 203 Maxwell Centre, Durban
  - 700 Medi Centre, Durban
  - Mount Edgecombe Medical Centre, Suite 15, Durban
  - Randles Rd Medical Centre, Durban
  - 1644 Starling Street, Johannesburg
  - Centre for Diabetes & Endocrinology, Johannesburg
  - DJW Navorsing, Johannesburg
  - Melrose Arch, Johannesburg
  - Seva Sadan, Room 6, Johannesburg
  - Union Hospital, Room 209, Johannesburg
  - Wits Donald Gordon Clinical Trial Site, Johannesburg
  - Mercantile Hospital, Port Elizabeth
  - 122 Louis Pasteur Building, Pretoria
  - 456 Leyd Steer, Pretoria
  - Eastmed Medical Centre, Pretoria
  - GCT Trial Centre Jubilee, Jubilee Hospital, Pretoria
  - The Bay Hospital, Suite M5, Richards Bay
  - Helderberg Diabetes and Medical Centre, Somerset West
  - 14 Medgate Medical Centre, Umhlanga
- Ukraine (13):
  - Department of Endocrinology of Bukovina State Medical University, Chernivtsy
  - Institute of Problem of Endocrinological Pathology UAMS., Kharkiv
  - Kharkov Regional Clinical Hospital, Kharkiv
  - Bogomolets National Medical University, Kiev
  - Department of Endocrinology, Scientific Center of Radiation Medicine, Kiev
  - Komisarenko Institute of Endocrinology and Metabolism of UAMS, Kiev
  - Ukrainian Scientific and Practical Center of Endocrinology Surgery, Kiev
  - Lviv Regional Endocrinology Health Center, Lviv
  - Odessa State Medical University., Odesa
  - M.V. Sklifosovskiy Regional Clinical Hospital., Poltava
  - Semashko Republic Clinical Hospital, Simferopol
  - Reginal Clinical Endocrinological Health Center, Vinnitsa
  - Basin Clinical Hospital, Zaporizhya